CLINICAL TRIAL: NCT00046033
Title: A Phase II, Randomized, Open-Label Study Comparing Fixed-Dose Versus Concentration-Adjusted Lopinavir/Ritonavir Therapy in HIV-Infected Subjects on Salvage Therapy
Brief Title: Comparing Standard-Dose Versus Adjusted-Dose Lopinavir/Ritonavir Therapy in HIV-Infected Persons With Drug Resistance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5135
Record Dates: First submitted 2002-09-18; First posted 2002-09-19 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2005-05

CONDITIONS: HIV Infections
Keywords: Dose-Relationship, Drug; HIV Protease Inhibitors; Salvage Therapy; Viral Load; RNA, Viral; Drug Therapy, Combination
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; Ritonavir; Saquinavir; Tenofovir; amprenavir

INTERVENTIONS:
Drug: Lopinavir/ritonavir
Drug: Ritonavir
Drug: Saquinavir
Drug: Tenofovir disoproxil fumarate
Drug: Amprenavir

SUMMARY:
The purpose of this study is to see if adjusting the dose of lopinavir/ritonavir (LPV/r) has a better effect on lowering HIV viral load (the amount of HIV in the blood) compared to taking the standard FDA-approved LPV/r dose. This study will also compare the safety and tolerability of these two types of dosing.

DETAILED DESCRIPTION:
Antiretroviral drugs may fail to suppress HIV unless there are adequate amounts of those drugs in the blood. By monitoring the amounts of drugs in the blood and adjusting doses to achieve optimal drug concentrations, response to antiretroviral drugs may improve, especially in patients who have failed previous regimens. This study is designed to evaluate drug monitoring and dose adjustment of protease inhibitors (PIs) in heavily treatment-experienced patients.

Patients will be randomized to receive either a standard dose of LPV/r (Arm A) or a concentration-adjusted dose of LPV/r (Arm B). Concentration-adjusted dosing means that the dose of ritonavir or lopinavir may be increased based on the amount of lopinavir measured in the blood and the results of a drug resistance test. All patients start the study taking LPV/r, tenofovir disoproxil fumarate (TDF), 0 to 2 additional nucleoside reverse transcriptase inhibitors (NRTIs), and saquinavir (SQV) or amprenavir (APV). Only LPV/r, TDF, and SQV will be provided by the study. Other medications taken as part of the antiretroviral regimen must be obtained outside the study.

Patients in Arm A will take the usual approved dose of LPV/r for the first 24 weeks. At Week 24, patients with high viral loads will come to the clinic for a 12-hour LPV blood level measurement to see if the level of LPV needs to be increased. If it does, an additional capsule of ritonavir will be added to the regimen to boost the level of LPV.

Patients in Arm B will have a series of blood draws over a 12-hour period in the clinic, around 14 days after starting the study, to find out if their LPV level needs to be increased. If the LPV level needs to be raised, an additional capsule of ritonavir will be added to the regimen to boost the level of LPV. Patients who had their ritonavir dose adjusted will return to have another 12-hour blood draw around Week 5. If the LPV level still needs to be changed, an additional capsule of LPV/r will be added to the regimen. A third 12-hour blood draw will be performed around Week 8 if a second dose adjustment was necessary.

During the study, patients will visit the clinic weekly through Week 6, again at Week 8, then every 4 weeks thereafter through Week 32. Patients will have blood drawn at certain visits to test for LPV level, viral load, CD4 count, fasting lipids and glucose, and drug resistance.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infection
* Viral load >= 5000 copies/ml within 45 days prior to study entry
* Documented reduction in LPV sensitivity based on results obtained within 45 days prior to study entry
* Prior experience with 2 or more NRTIs for at least 6 months each
* At least 12 weeks of stable antiretroviral treatment that includes at least one PI prior to study entry and may include TDF and/or T-20 for 8 weeks or more immediately prior to study entry
* Negative pregnancy test within 14 days prior to study entry
* Agree not to become pregnant or to impregnate and to use an acceptable form of contraception while receiving study drugs and for 4 weeks after stopping study drugs

Exclusion Criteria:

* Pregnant or breast-feeding.
* Certain drugs within 14 days prior to study entry
* Nonnucleoside reverse transcriptase inhibitors (NNRTIs) within 14 days prior to study entry
* History of intolerance to LPV/r, RTV, or TDF and/or their components
* Drug or alcohol use that, in the opinion of the investigator, would interfere with the study
* Require therapy and/or hospitalization due to a serious infection or medical illness that is potentially life-threatening within 14 days prior to study entry
* Any condition that, in the opinion of the investigator, would compromise ability to participate in the study
* Unexplained fever for 7 consecutive days or chronic diarrhea within 30 days prior to study entry
* Cancer requiring chemotherapy
* Any immune system drugs, HIV vaccine, or other experimental therapy within 30 days prior to study entry
* Plan to use any PI other than APV, SQV, or LPV/r in the initial study treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118
Dates: Primary Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah McMahon, M.D., Study Chair — University of Pittsburgh
Locations (6):
- United States (6):
  - Univ of Miami, Miami, Florida
  - Univ of Hawaii, Honolulu, Hawaii
  - NYU/Bellevue, New York, New York
  - Case Western Reserve Univ, Cleveland, Ohio
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Univ of Texas, Galveston, Galveston, Texas

REFERENCES:
- [Background] Durant J, Clevenbergh P, Garraffo R, Halfon P, Icard S, Del Giudice P, Montagne N, Schapiro JM, Dellamonica P. Importance of protease inhibitor plasma levels in HIV-infected patients treated with genotypic-guided therapy: pharmacological data from the Viradapt Study. AIDS. 2000 Jul 7;14(10):1333-9. doi: 10.1097/00002030-200007070-00005. PMID 10930147
- [Background] Kilby JM, Hill A, Buss N. The effect of ritonavir on saquinavir plasma concentration is independent of ritonavir dosage: combined analysis of pharmacokinetic data from 97 subjects. HIV Med. 2002 Apr;3(2):97-104. doi: 10.1046/j.1468-1293.2002.00090.x. PMID 12010356
- [Background] Veldkamp AI, van Heeswijk RP, Mulder JW, Meenhorst PL, Schreij G, van der Geest S, Lange JM, Beijnen JH, Hoetelmans RM. Steady-state pharmacokinetics of twice-daily dosing of saquinavir plus ritonavir in HIV-1-infected individuals. J Acquir Immune Defic Syndr. 2001 Aug 1;27(4):344-9. doi: 10.1097/00126334-200108010-00004. PMID 11468422